CLINICAL TRIAL: NCT04496726
Title: A Proof-of-concept, Feasibility Study to Investigate the Effect of Cranberry and Quillaia Extract Type II on Symptoms in Women With Uncomplicated Urinary Tract Infection and to Study the Modulation of the Urinary and Gut Microbiome Pre- and Post-antibiotic Use
Brief Title: Cranberry and Quillaja on Symptoms of Uncomplicated UTI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure to recruit
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Urobiome Therapeutics (Unknown); St. Joseph's Health Care London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00043294
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Urinary Tract Infections; UTI; UTI - Lower Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: Open label, single site, single group prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cranberry and Quillaja (Experimental): one 450mg cranberry capsule and one 50mg quillaja capsule in the morning and evening for 14 days.
  Interventions: Other: Pacran and Sapnov P quillaja

INTERVENTIONS:
Other: Pacran and Sapnov P quillaja — Cranberry (450 mg) and quillaja (50 mg) capsules taken orally twice daily (morning and evening) for a total daily dose of 900 mg cranberry and 100 mg quillaja for 14 days. Nitrofurantoin 100 mg taken orally twice daily for five days as a rescue medication if symptoms do not subside.
  Other Names: Cranberry; Quillaja; Pacran; Naturex; Sapnov P; Quillaia extract type II

SUMMARY:
This study will investigate the effects of cranberry and quillaja capsules on symptoms of uncomplicated urinary tract infections.

DETAILED DESCRIPTION:
Urinary tract infection (UTI) is one of the most common bacterial infections in humans and it disproportionately affects women. Currently there are only a few alternatives to antibiotics for treatment of UTI. Although symptomatic relief occurs more quickly in women treated with oral antibiotics for uncomplicated UTIs, patients appear to successfully resolve their UTI without antibiotic therapy. While antibiotics are the mainstay of therapy, there are growing concerns about collateral effects impacting healthy microbiomes and anti-bacterial resistance patterns. Recent estimates from the CDC indicate that more than 2.8 million antibiotic-resistant infections occur in the U.S. each year, and more than 35,000 people die as a result.

The proposed research fills a key knowledge gap that will be critical in determining the role of a non-antibiotic substance with the potential to treat UTIs by modulating the urinary and gut microbiome to restore health and minimize the reliance on traditional antibiotic therapy while also preventing antibiotic resistance. In addition, this study will provide early evidence of the short-term symptom and urinary and gut microbiome changes following ingestion of two botanical food substances (cranberry and quillaja) that have the potential for beneficial effects on the microbiome and UTI symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-menopausal women 18 years and over
2. Presenting with typical symptoms of an uncomplicated UTI
3. Positive leukocyte or nitrite on in-office urine dipstick confirmed
4. Able to swallow capsules
5. Willing and able to fill out/ answer questionnaires and comply with the study requirement
6. Willing to initiate clinically prescribed antibiotic therapy (typically 5-day antibiotic).
7. Provided written informed consent
8. BMI >17.5kg m2 and <35kg m2

Exclusion Criteria:

1. Regular use of Vaccinium containing products (e.g. all forms of blueberries, cranberries, bilberry, lingonberry etc. i.e. fruit, dried fruit, pills, juices or supplements) within 28 days of Day 1,
2. Allergy to cranberry, tree bark, or quillaja.
3. Use of any antibacterial supplements or products, that in the opinion of the Medical Investigator may interfere with the study outcomes, within 28 days of Day 1
4. A history of >5 UTIs in the last 6 months (confirmed by self-report or health professional)
5. Use of antibiotics or antibiotics for prophylaxis to treat a UTI within 28 days of Day 1
6. Women of child bearing potential not willing to use adequate and effective methods of contraception throughout the study, in the opinion of the Investigator
7. Positive urine dipstick pregnancy test at screening on Day 1, currently pregnant and/or breastfeeding
8. History of an adverse reaction or known hypersensitivity or suspected allergy to the investigational product ingredients
9. History of pyelonephritis or reflux
10. Presence of an intermittent or indwelling urinary catheter
11. Anatomical abnormalities of the urinary tract (self-reported)
12. History of or known clinically significant renal or urological disease (self-reported), at the discretion of the investigator
13. History of or known clinically significant cardiac disease, at the discretion of the investigator
14. History of or known clinically significant liver disease, at the discretion of the investigator
15. History of or known clinically significant gastrointestinal disease, at the discretion of the investigator
16. History of or known metabolic disorder or diabetes
17. History of or known incomplete emptying of bladder
18. History or presence of alcohol or illicit drug abuse, any surgical history, clinical condition or organ dysfunction that in the opinion of the Medical Investigator may affect the participant's ability to participate in the study or the study results
19. Currently hospitalized or any planned hospitalizations within the study period.
20. Immunocompromised participants or participants receiving immunosuppressive medication
21. Currently taking warfarin or has received Warfarin within 28 days of Day 1
22. Received an investigational drug within 28 days of Day 1 (pills, juices or supplements)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Urinary Tract Infection Symptoms Assessment Questionnaire (UTISA) | 14 days
  This questionnaire assesses the degree of symptoms and bother on a scale of 0 to 3, and has 3 domains of urinary regularity, problems with urination and pain associated with urination. The fourth domain includes the presence of hematuria. Subjects will complete the UTISA questionnaire every day for 14 days.
Time to UTI antibiotic initiation | 14 days
  This will be assessed using study form, UTI Comfort Measure Assessment. Subjects will have access to a clinically prescribed UTI antibiotic, nitrofurantoin 100mg. Subjects will be asked to record each day their intake of any antibiotic during the study period.

SECONDARY OUTCOMES:
Microbiome changes prior to and post antibiotic initiation | 14 days
  This outcome measure can only be assessed for those participants that require antibiotic initiation. Changes in the entire bacterial community prior to and post antibiotic use will be assessed in the lab from faecal and urine samples collected by the participant. The microbes may vary by participant and the study will be looking at which ones present themselves in each case. Units of measure via culture are colony forming units per g (cfu/g).

CONTACTS AND LOCATIONS:
Overall Officials: Blayne Welk, MD, Principal Investigator — St. Joseph's Healthcare London
Locations (1):
- St. Joseph's Health Care London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Falagas ME, Kotsantis IK, Vouloumanou EK, Rafailidis PI. Antibiotics versus placebo in the treatment of women with uncomplicated cystitis: a meta-analysis of randomized controlled trials. J Infect. 2009 Feb;58(2):91-102. doi: 10.1016/j.jinf.2008.12.009. Epub 2009 Feb 4. PMID 19195714
- [Background] Pappas E, Schaich KM. Phytochemicals of cranberries and cranberry products: characterization, potential health effects, and processing stability. Crit Rev Food Sci Nutr. 2009 Oct;49(9):741-81. doi: 10.1080/10408390802145377. PMID 20443158
- [Background] Howell AB, Reed JD, Krueger CG, Winterbottom R, Cunningham DG, Leahy M. A-type cranberry proanthocyanidins and uropathogenic bacterial anti-adhesion activity. Phytochemistry. 2005 Sep;66(18):2281-91. doi: 10.1016/j.phytochem.2005.05.022. PMID 16055161
- [Background] Vostalova J, Vidlar A, Simanek V, Galandakova A, Kosina P, Vacek J, Vrbkova J, Zimmermann BF, Ulrichova J, Student V. Are High Proanthocyanidins Key to Cranberry Efficacy in the Prevention of Recurrent Urinary Tract Infection? Phytother Res. 2015 Oct;29(10):1559-67. doi: 10.1002/ptr.5427. Epub 2015 Aug 13. PMID 26268913
- [Background] Sarkhel S. Evaluation of the anti-inflammatory activities of Quillaja saponaria Mol. saponin extract in mice. Toxicol Rep. 2015 Dec 1;3:1-3. doi: 10.1016/j.toxrep.2015.11.006. eCollection 2016. PMID 28959520
- [Background] Fleck JD, Betti AH, da Silva FP, Troian EA, Olivaro C, Ferreira F, Verza SG. Saponins from Quillaja saponaria and Quillaja brasiliensis: Particular Chemical Characteristics and Biological Activities. Molecules. 2019 Jan 4;24(1):171. doi: 10.3390/molecules24010171. PMID 30621160
- [Background] den Brok MH, Bull C, Wassink M, de Graaf AM, Wagenaars JA, Minderman M, Thakur M, Amigorena S, Rijke EO, Schrier CC, Adema GJ. Saponin-based adjuvants induce cross-presentation in dendritic cells by intracellular lipid body formation. Nat Commun. 2016 Nov 7;7:13324. doi: 10.1038/ncomms13324. PMID 27819292
- [Background] Southworth E, Hochstedler B, Price TK, Joyce C, Wolfe AJ, Mueller ER. A Cross-sectional Pilot Cohort Study Comparing Standard Urine Collection to the Peezy Midstream Device for Research Studies Involving Women. Female Pelvic Med Reconstr Surg. 2019 Mar/Apr;25(2):e28-e33. doi: 10.1097/SPV.0000000000000693. PMID 30807432
- See also: A Randomized, Double Blind, Controlled, Dose Dependent Clinical Trial to Evaluate the Efficacy of a Proanthocyanidin Standardized Whole Cranberry (Vaccinium macrocarpon) Powder on Infections of the Urinary Tract. Current Bioactive Compounds — https://www.researchgate.net/publication/233632623_A_Randomized_Double_Blind_Controlled_Dose_Dependent_Clinical_Trial_to_Evaluate_the_Efficacy_of_a_Proanthocyanidin_Standardized_Whole_Cranberry_Vaccinium_macrocarpon_Powder_on_Infections_of_the_Urinary
- See also: Quillaja Saponaria Extract; Exempt from the Requirement of a Tolerance — https://www.federalregister.gov/documents/2007/08/01/E7-14894/quillaja-saponaria-extract-exemption-from-the-requirement-of-a-tolerance